CLINICAL TRIAL: NCT05878210
Title: A Phase IV Study to Evaluate the SUBLOCADE Treatment Exit Strategy
Brief Title: Evaluating the SUBLOCADE Treatment Exit Strategy
Status: Completed | Type: Observational
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: INDV-6000-407
Record Dates: First submitted 2023-05-04; First posted 2023-05-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
Keywords: Medicine for Opioid Use Disorder (MOUD)
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to observe and assess the successful taper and opioid withdrawal experience after participants stop receiving SUBLOCADE because their healthcare provider determines their disease symptoms have been controlled for at least 9 months and they, together with their healthcare provider, plan to discontinue MOUD.

DETAILED DESCRIPTION:
This is a Phase IV, observational, multicentre, open-label, study in participants with a history of OUD, who have been on SUBLOCADE treatment for at least 12 injections, have had disease symptoms controlled for at least 9 months in the opinion of the healthcare provider, and both healthcare provider and participant plan to discontinue MOUD treatment.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria:

* The participant, together with their healthcare provider (the investigator), have previously determined that it is appropriate to stop MOUD treatment, and the participant meets the following criteria:

  * Has been treated with at least 12 injections of SUBLOCADE.
  * In the opinion of the investigator, has had their OUD symptoms (ie, overdose, illicit/nonmedical use, withdrawal) controlled for at least 9 months.
  * In the opinion of the investigator, has had any other substance use disorder (excluding alcohol, nicotine, or cannabis) symptoms controlled for at least 9 months.
* Is willing to complete the Baseline Visit 4 to 8 weeks after the last dose of SUBLOCADE.
* Has signed the ICF and is 18 years of age or older.
* Is not currently using opioids to treat a diagnosis other than OUD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a history of OUD, who have been on SUBLOCADE treatment for at least 12 injections, have disease symptoms controlled for at least 9 months in the opinion of the healthcare provider, and discontinue SUBLOCADE treatment.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Rate of successful taper by the end of 6-month follow-up. | 6 months
  * Successful taper is defined as no consistent self-reported illicit/nonmedical opioid use and not restarting long-term MOUD treatment due to opioid withdrawal or illicit/nonmedical opioid use during follow up.
  * Consistent self-reported illicit/nonmedical opioid use is defined as self-reported 4 consecutive use weeks (ie, weeks with at least 1 day of illicit/nonmedical opioid use per week) or 7 consecutive days of illicit/nonmedical opioid use.

SECONDARY OUTCOMES:
Key secondary - At each given month, for participants not restarting MOUD and not consistently using illicit/nonmedical opioid up to the start of that month: | 6 months
  Average clinical experience score (range: 0 to 4 with higher score = worse outcome) on opioid withdrawal severity during the past month
Participants restarting MOUD (yes/no) during study follow-up | 6 months
  Yes/No
Participants who reported withdrawal symptoms (yes/no) during the past month | 6 months
  Yes/No
Participants who used ancillary medications to treat opioid withdrawal symptoms (yes/no) during the past month | 6 months
  Yes/No
Participants who used rescue MOUD (yes/no) to treat opioid withdrawal symptoms during the past month | 6 months
  Yes/No
Participants who had self-reported illicit/nonmedical opioid use (yes/no) during the past month | 6 months
  Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: (804) 594-4488, Study Director — Indivior Inc.
Locations (2):
- Comprehensive Addiction Medicine, Portland, Maine, United States
- Savera Medical Centre, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No